CLINICAL TRIAL: NCT04813107
Title: A Phase I/II Open-Label Multicenter Study to Evaluate the Safety and Efficacy of Oral APL-1202 in Combination With Tislelizumab Compared to Tislelizumab Alone as Neoadjuvant Therapy in Patients With Muscle Invasive Bladder Cancer (MIBC)
Brief Title: A Study to Evaluate the Safety and Efficacy of Oral APL-1202 in Combination With Tislelizumab Compared to Tislelizumab Alone as Neoadjuvant Therapy in Patients With Muscle Invasive Bladder Cancer
Acronym: ANTICIPATE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Yahong Meditech Co., Ltd aka Asieris (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YHGT-NP-01
Record Dates: First submitted 2021-03-21; First posted 2021-03-24 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Muscle Invasive Bladder Cancer
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- APL-1202 in combination with tislelizumab (Active Comparator)
  Interventions: Drug: APL-1202 in combination with tislelizumab
- Tislelizumab alone (Placebo Comparator)
  Interventions: Drug: Tislelizumab alone

INTERVENTIONS:
Drug: APL-1202 in combination with tislelizumab — For those assigned to this group (1), each patient will receive 3 cycles of treatment prior to RC and each cycle is 3 weeks. On day 1 of each cycle, a single dose of 200 mg tislelizumab will be administered intravenously. APL-1202 will be administered orally TID daily for 3 weeks at the RP2D defined from Phase I.
  Arms: APL-1202 in combination with tislelizumab
Drug: Tislelizumab alone — For patients assigned to this group (2), each patient will receive 3 cycles of treatments with a single dose of 200 mg tislelizumab administered on day 1 of each cycle, followed by RC.
  Arms: Tislelizumab alone

SUMMARY:
This trial is designed to evaluate the safety, efficacy, and biomarker response of APL-1202 in combination with tislelizumab as neoadjuvant therapy for patients with MIBC who are cisplatin ineligible or refuse cisplatin-based chemotherapy.

DETAILED DESCRIPTION:
This trial is an open-label, multi-center clinical study consisting of two periods: Phase Ⅰ and Phase Ⅱ. Phase I is a dose escalation study to determine MTD (maximum tolerated dose) and/or RP2D. Phase II is an expanded proof of concept (POC) study to evaluate the safety and efficacy of APL-1202 in combination with tislelizumab compared to tislelizumab alone as neoadjuvant therapy for MIBC as measured by pCR.

Phase Ⅰ and Phase Ⅱ both are divided into 3 periods: screening period, neoadjuvant therapy and follow-up period:

* The screening period is up to 4 weeks before the first doses of study treatments.
* During the neoadjuvant therapy, each patient will receive the combined treatment of tislelizumab and APL-1202 or tislelizumab alone, every 21 days as a dosing cycle for a total of 3 cycles of treatment prior to radical cystectomy.
* The follow-up period includes a safety follow-up at 4 weeks after radical cystectomy.

Phase Ⅰ: Dose-Escalation The dose escalation phase will assess the safety, tolerability, and pharmacokinetics of APL-1202 in combination with tislelizumab in MIBC patients. Results from this period will determine the RP2D of APL-1202 in combination with tislelizumab as neoadjuvant therapy for MIBC.

Patients enrolled in this phase must meet the following criteria: those with newly diagnosed MIBC for whom RC is planned, and who are cisplatin ineligible or refuse to receive cisplatin based neoadjuvant chemotherapy, and with calculated CrCl ≥ 50 mL/min (by Cockcroft-Gault equation).

A standard 3+3 dose-escalation design will be used. The dose of APL-1202 will start at 375 mg (125 mg, TID) and increase sequentially to 750 mg (250 mg, TID) and 1,125 mg (375 mg, TID). For more information on the dose escalation design, please see the Dose Escalation Criteria section.

Table 1: Dose-Escalation plan

Dose Level Tislelizumab APL-1202 Patients (n)

1. 200 mg, IV, Q3w 125 mg, PO, TID ≥ 3
2. 200 mg, IV, Q3w 250 mg, PO, TID ≥ 3
3. 200 mg, IV, Q3w 375 mg, PO, TID ≥ 3 Patients will be assigned to one of three APL-1202 dose levels. Each patient will receive 3 cycles of treatment prior to RC and each cycle is 3 weeks. On day 1 of each cycle, a single dose of 200 mg tislelizumab will be administered intravenously and APL-1202 will be administered orally TID daily for 3 weeks. If the dose level 1 is determined to be safe and tolerable, 3 patients will be enrolled to Dose Level 2 and will receive their treatments in 3-week treatment cycles and safety will be assessed. This process is repeated one more time for the Dose Level 3.

The DLT observation window for any dose level will be treatment cycle 1 (1-21 days).

Patients who do not complete the DLT observation period (cycle 1) will be replaced unless the discontinuation of treatment is DLT-related.

DLT assessment will be performed during the first cycle (1-21 days) of study treatments. An evaluable patient is defined as a patient who has received at least 75% of planned APL-1202 doses during the first cycle of treatment and completed all the safety evaluations required for the first cycle, or any patient who has DLT during the first cycle. If a patient receives less than 75% of planned APL-1202 doses during the first cycle or withdraws from the study due to reasons other than DLT, the patient will be replaced.

There will be no intra-patient dose escalation. A patient will receive treatments of cycle 2 and cycle 3 or until unacceptable toxicity, disease progression, or discontinuation for any other reason.

Phase Ⅱ: Proof of Concept (POC) The primary objective of this phase is to evaluate the safety and efficacy of APL-1202 in combination with tislelizumab compared to tislelizumab alone as neoadjuvant therapy for MIBC as measured by pathologic complete response (pCR).

Patients enrolled in this phase must meet the following criteria: those with newly diagnosed MIBC for whom RC is planned, and who are cisplatin ineligible or refuse to receive cisplatin based neoadjuvant chemotherapy.

As shown in Figure 1 below, eligible patients will be randomly assigned to group 1 or group 2, with PD-L1expression level as a stratification factor. For those assigned to group 1, each patient will receive 3 cycles of treatment prior to RC and each cycle is 3 weeks. On day 1 of each cycle, a single dose of 200 mg tislelizumab will be administered intravenously. APL-1202 will be administered orally TID daily for 3 weeks at the RP2D defined from Phase I. For patients assigned to group 2, each patient will receive 3 cycles of treatments with a single dose of 200 mg tislelizumab administered on day 1 of each cycle, followed by RC. A patient will stay on treatment until completion of planned treatments, unacceptable toxicity, disease progression, or discontinuation for any other reason.

In this period, patients with renal function with calculated CrCl ≥ 30 mL/min (by Cockcroft-Gault equation) will be recruited. if patients with CrCl ≥ 50 mL/min, start dose of APL-1202 is recommended to be RP2D defined from Phase I; for patients with CrCl 30-50 mL/min, the dose of APL-1202 is recommended to be reduced by 1 dose level from RP2D defined from Phase I (from 1125 mg/day to 750 mg/day, or from 750 mg/day to 375 mg/day).

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Age ≥ 18 years.
3. Histopathologically confirmed transitional cell carcinoma of the bladder. Patients with mixed histologies are required to have a dominant (i.e. > 50%) transitional cell pattern.
4. Radical cystectomy is planned (according to local guidelines).
5. Patients who refuse neoadjuvant cisplatin based chemotherapy or in whom neoadjuvant cisplatin based therapy is contraindicated. Contraindications to cisplatin is defined by meeting at least one of the following criteria:

   * Impaired renal function with calculated CrCl 30 to 59 mL/min (by Cockcroft-Gault equation).
   * Eastern Cooperative Oncology Group (ECOG) Performance Status 2.
   * CTCAE v.5 Grade ≥2 audiometric hearing loss.
   * In the clinical judgement of the investigator, potential adverse effects from cisplatin-based neoadjuvant chemotherapy outweighs its benefits.
6. Clinical stage T2-T4a N0 M0 disease by CT (or MRI) (within 4 weeks of randomization).
7. Residual disease after transurethral resection of bladder (TURB) (surgical opinion, cystoscopy or radiological presence).
8. Availability of representative formalin-fixed paraffin-embedded (FFPE) tumor specimens or unstained slides, with an associated pathology report, and determined to be evaluable for tumor PD-L1 expression prior to study enrollment;
9. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
10. Adequate hematologic and end-organ functions:

    * Hemoglobin > 9.0 g/dL;
    * Absolute neutrophil count (ANC) > 1.5×109 /L;
    * Platelet count > 100×109 /L;
    * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN).
    * Aspartate aminotransferase (AST) /alanine aminotransferase (ALT) ≤ 2.5 x institutional upper limit of normal ULN.
    * CrCl (calculated using Cockcroft-Gault equation) ≥ 30 mL/min (calculated CrCl ≥ 50 mL/min in Phase Ⅰ: Dose-Escalation).
    * INR < 1.5. This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose.
11. Female patients should be surgically sterilized or post-menopausal or must agree to take effective contraceptive measures during the treatment. Male patients must be surgically sterilized or must agree to take effective contraceptive measures during treatment. Patients must continue to take contraceptive measures for 3 months after the investigational therapy was completed.

Exclusion Criteria:

1. Previous systemic therapy for bladder cancer.
2. Malignancies other than urothelial bladder cancer within 5 years prior to cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ of breast treated surgically with curative intent).
3. Evidence of measurable nodal or metastatic disease.
4. Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including significant liver disease (such as cirrhosis, uncontrolled major seizure disorder, or superior vena cava syndrome).
5. Pregnant female patients. All female patients with a positive pregnancy test within 2 weeks prior to the first dose of study treatment will be excluded from the study.
6. Significant cardiovascular disease, such as New York Heart Association cardiac disease (more than Class II), myocardial infarction within 3 months prior to enrollment, unstable arrhythmias, or unstable angina.
7. Severe infections within 4 weeks prior to enrollment in the study including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
8. Major surgical procedure within 4 weeks prior to enrollment or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis.
9. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
10. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the tislelizumab or APL-1202 formulation.
11. History of autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.
12. History of autoimmune-related hypothyroidism, unless on a stable dose of thyroid-replacement hormone.
13. History of idiopathic pulmonary fibrosis.
14. Uncontrolled Type 1 diabetes mellitus.
15. Uncontrolled hypercalcemia (> 1.5 mmol/L ionized calcium or calcium > 12 mg/dL or corrected serum calcium > ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab.
16. Prior allogeneic stem cell or solid organ transplantation.
17. Positive test for HIV.
18. Uncontrolled hepatitis infection.
19. Active tuberculosis.
20. Optic nerve disorders or with a history of optic nerve disorders.
21. Cataract or with a history of cataract.
22. Prior treatment with anti-programmed death-1 (PD-1), or anti-PD-L1 therapeutic antibody or pathway-targeting agents.
23. Patients taking regular oral steroids, above the allowed limit of 10 mg/day methylprednisolone/prednisone or analogues, for any reason. Patients must not have had steroids for 4 weeks prior to study entry.
24. Administration of vaccine within 4 weeks prior to enrollment or anticipation that such a vaccine will be required during the study.
25. Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 4 weeks prior to enrollment.
26. Treatment with systemic immunostimulatory agents within 4 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2021-12-28 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AE) and serious adverse events (SAE). | 9 weeks
  Adverse events (AE) and serious adverse events (SAE) in Phase Ⅰ(Dose-Escalation)
The RP2D of APL-1202 in combination with tislelizumab. | 9 weeks
  The RP2D of APL-1202 in combination with tislelizumab in Phase Ⅰ(Dose-Escalation)
The rate of pathologic complete response (pCR) in Phase 2. | 26 months
  Pathological complete response (pCR) is defined as no microscopic evidence of residual disease in the bladder based on histological evaluation of the resected bladder specimen collected during cystectomy.

SECONDARY OUTCOMES:
Radiological response (RR). | 26 months
  CT or MRI scan taken at screening and pre-radical cystectomy visits. Response will be evaluated using standard RECIST 1.1 criteria.
Cmax | 26 months
  PK parameters of APL-1202 expressed as Cmax when administered concurrently with tislelizumab.
Tmax | 26 months
  PK parameters of APL-1202 expressed as Tmax when administered concurrently with tislelizumab.
t1/2 | 26 months
  PK parameters of APL-1202 expressed as t1/2 when administered concurrently with tislelizumab.
AUC | 26 months
  PK parameters of APL-1202 expressed as AUC when administered concurrently with tislelizumab.
Cumulative amount in urinary excretion (Ae) | 26 months
  PK parameters of APL-1202 expressed as Ae when administered concurrently with tislelizumab.
cumulative fraction of dose in urinary excretion (Ae%) | 26 months
  PK parameters of APL-1202 expressed as Ae% when administered concurrently with tislelizumab.
Tumor mutation burdens (TMB) in pre- and post-treatment plasma ctDNA (circulating tumor DNA). | 26 months
  Plasma circulating tumor DNA (ctDNA) were extracted from the patients before and after treatment; somatic mutations were detected by targeted region sequencing. Tumor mutation burdens (TMB) was calculated by mutations per million sequenced bases.
Tumor mutation burdens (TMB) in pre- and post-treatment urine cfDNA (cell free DNA). | 26 months
  Urine cell free DNA (cfDNA) were extracted from the patients before and after treatment; somatic mutations were detected by targeted region sequencing. Tumor mutation burdens (TMB) was calculated by mutations per million sequenced bases.
Tumor mutation burdens (TMB) in pre- and post-treatment tumor tissues. | 26 months
  Tumor tissue FFPE slides were collected from the patients before and after treatment. DNA was extracted from the FFPE slides. Somatic mutations were detected by targeted region sequencing. Tumor mutation burdens (TMB) was calculated by mutations per million sequenced bases.
PD-L1 protein expression levels in pre- and post-treatment tumor tissues. | 26 months
  Tumor tissue FFPE slides were collected from the patients before and after treatment. PD-L1 protein expression levels were evaluated by IHC (immunohistochemistry, VENTANA PD-L1/SP263 Assay).

CONTACTS AND LOCATIONS:
Locations (2):
- Mount Sinai Medical Center, New York, New York, United States
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No